CLINICAL TRIAL: NCT02552368
Title: A Brain Computer Interface and Brain-Controlled Stroke Rehabilitation Method Utilizing Electroencephalography in Hemiparetic and Hemiplegic Stroke Patients to Achieve Thought Control of Machines and a Better Understanding of Brain Function
Brief Title: Treatment of Chronic Stroke With IpsiHand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201021771
Record Dates: First submitted 2015-08-22; First posted 2015-09-17 (Estimated); Results first posted 2018-09-17 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Stroke
Keywords: Stroke Rehabilitation; BCI; Stroke; Upper Extremity Rehabilitation; paresis; hemiparesis
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IpsiHand (Experimental): IpsiHand is a device which includes a robotic glove that you wear on your hand and a headset that you wear on your head. The headset picks up your thoughts and sends them to the robotic glove, to control opening and closing of your hand.
  Interventions: Device: IpsiHand Device

INTERVENTIONS:
Device: IpsiHand Device — Once a participant has completed (3) EEG Signal Screens and (2) separate set of baseline measurements, the IpsiHand BCI Device is provided to participants to use a minimum of (5) out of (7) days a week for a total duration of 12 weeks. Participants are seen bi-weekly throughout the duration of the trial to assess affected upper extremity and assess functional impact. At the completion of 12 weeks of device use, the participants complete a set of measurements to assess function of the affected upper extremity.

SUMMARY:
The ultimate goal of this project is to develop a functioning and clinically feasible method for restoring function to motor-impaired stroke survivors. This ultimate goal will be approached through two different means. The first method is to develop a functioning brain-computer interface that operates based on cortical activity ipsilateral to an intended movement on the motor-impaired side of the body. And secondly, to develop new methods of rehabilitation that involve stimulating peripheral muscles based upon cortical activity ipsilateral to intended movements. Finally, the study seeks to assess changes in functional connectivity as a result of using a BCI device.

DETAILED DESCRIPTION:
This study will be carried out in two phases designed to achieve the objectives described above. The first phase will determine the feasibility of recording ipsilateral (contralesional) motor commands and use the signals to control a computer. This phase will involve recording EEG signals during the performance of real and imagined motor movements of both the impaired and non-impaired hand in stroke survivors. After recording the signals and analyzing the data, the signals will be used to try to control a cursor on a computer screen or a robotic hand. The second phase of the study will determine if the BCI system can be used to impact rehabilitation. Motor commands would be performed as in phase 1 to determine the accompanying EEG signals. The EEG signals would then be used to control stimulation of the impaired limb. Rehabilitation would be assessed by examining changes in commonly used functional motor scores.

The ultimate goal of this project is to develop a functioning and clinically feasible method for restoring function to motor-impaired stroke survivors. This ultimate goal will be approached through two different means. The first method is to develop a functioning brain-computer interface that operates based on cortical activity ipsilateral to an intended movement on the motor-impaired side of the body. And secondly, to develop new methods of rehabilitation that involve stimulating peripheral muscles based upon cortical activity ipsilateral to intended movements. Finally, the study seeks to assess changes in functional connectivity as a result of using a BCI device.

ELIGIBILITY:
Inclusion Criteria:

* 6 months post stroke
* Modified Ashworth Scale of 1+ or less of elbow flexion in the affected upper extremity
* Short Blessed Test Score of 8 or less
* Unstructured Mesulam with 2 or less omissions

Exclusion Criteria:

* Dementia
* Severe spasticity in affected upper extremity
* Unilateral Visual Inattention (neglect)
* Contracture(s) in the affected upper extremity
* Botox injections administered within 9 months
* Aphasia which limits effective communication

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-08; Primary Completion 2015-11-30 (Actual); Study Completion 2015-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thy Huskey, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Bundy DT, Souders L, Baranyai K, Leonard L, Schalk G, Coker R, Moran DW, Huskey T, Leuthardt EC. Contralesional Brain-Computer Interface Control of a Powered Exoskeleton for Motor Recovery in Chronic Stroke Survivors. Stroke. 2017 Jul;48(7):1908-1915. doi: 10.1161/STROKEAHA.116.016304. Epub 2017 May 26. PMID 28550098

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IpsiHand
Started | 23
Completed | 10
Not Completed | 13

BASELINE CHARACTERISTICS:
Groups:
- Experimental: IpsiHand is a device which includes a robotic glove that you wear on your hand and a headset that you wear on your head. The headset picks up your thoughts and sends them to the robotic glove, to control opening and closing of your hand.
  IpsiHand Device: Once a participant has completed (3) EEG Signal Screens and (2) separate set of baseline measurements, the IpsiHand BCI Device is provided to participants to use a minimum of (5) out of (7) days a week for a total duration of 12 weeks. Participants are seen bi-weekly throughout the duration of the trial to assess affected upper extremity and assess functional impact. At the completion of 12 weeks of device use, the participants complete a set of measurements to assess function of the affected upper extremity.
Arm/Group | Experimental
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Action Research Arm Test (ARAT) Score
Description: The Action Research Arm Test (ARAT) is an evaluative measure to assess specific changes in limb function among individuals who sustained cortical damage resulting in hemiplegia (Lyle, 1981). It assesses a client's ability to handle objects differing in size, weight and shape and therefore can be considered to be an arm-specific measure of activity limitation (Platz, Pinkowski, Kim, di Bella, & Johnson, 2005).
  The ARAT's is a 19 item measure divided into 4 sub-tests (grasp, grip, pinch, and gross arm movement). Performance on each item is rated on a 4-point ordinal scale ranging from:
  3) Performs test normally 2) Completes test, but takes abnormally long or has great difficulty
  1) Performs test partially 0) Can perform no part of test
  The maximum score achievable on this measure is 57 points.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Change in ARAT From Baseline to 12 Weeks of BCI Device Use: IpsiHand is a device which includes a robotic glove that you wear on your hand and a headset that you wear on your head. The headset picks up your thoughts and sends them to the robotic glove, to control opening and closing of your hand.
Arm/Group | Change in ARAT From Baseline to 12 Weeks of BCI Device Use
Number analyzed (Participants) | 10
units on a scale | 6.2 (4.4)
Statistical Analysis 1: Comparison: Change in ARAT From Baseline to 12 Weeks of BCI Device Use; Test type: Superiority; p = 0.002, Paired t-Test

2. Secondary Outcome: Canadian Occupational Performance Measure (COPM)
Description: The COPM is an evidence-based outcome measure designed to capture a client's self-perception of performance in 5 patient-identified tasks over time. Patients identified 5 functional activities that they wanted to perform more independently or with greater ease. COPM measurements consisted of a semi-structured interview in which patients rated their performance & satisfaction with each activity on an ordinal scale from 1 to 10. A performance score of 1 indicated they are unable to perform identified task, & a score of 10 indicates they are able to complete the functional task as easy as prior to stroke. A satisfaction score of 1 indicated they were not satisfied at all to 10 indicating they are extremely satisfied with how they complete the identified functional task. Patients would rate (5) functional tasks for their performance and satisfaction. Scores were averaged between the scores from the 5 functional activities.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Change in COPM From Baseline to 12 Weeks of BCI Device Use: Ipsihand is a device that includes a robotic glove that you wear on your hand and a headset that you wear on your head. The headset picks up your thoughts and sends them to the robotic glove, to control opening and closing of your hand.
Arm/Group | Change in COPM From Baseline to 12 Weeks of BCI Device Use
Number analyzed (Participants) | 10
units on a scale
  Performance | 1.56 (1.70)
  Satisfaction | 1.54 (1.86)
Statistical Analysis 1: Comparison: Change in COPM From Baseline to 12 Weeks of BCI Device Use; Signed-Rank Test for Performance COPM between Baseline and 12 weeks; Test type: Superiority; p = 0.022, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Change in COPM From Baseline to 12 Weeks of BCI Device Use; Signed-Rank Test for Satisfaction COPM between Baseline and 12 weeks; Test type: Superiority; p = 0.031, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Groups:
- Chronic Stroke Survivors: All adverse events were monitored throughout the study completion, an average of 2 years with no events reported.
Arm/Group | Chronic Stroke Survivors
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No